CLINICAL TRIAL: NCT01278407
Title: A Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled Study of E2020 in Patients With Dementia With Lewy Bodies (DLB), Followed by a Long-term Extension Phase
Brief Title: A Study of E2020 in Patients With Dementia With Lewy Bodies (DLB), Followed by a Long-term Extension Phase
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E2020-J081-341
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Results first posted 2015-11-30 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2015-12

CONDITIONS: Dementia With Lewy Bodies (DLB)
Keywords: DLB; Dementia with Lewy bodies; Lewy Body Disease; Dementia; E2020; Donepezil; Aricept
MeSH Terms: conditions — Lewy Body Disease; Dementia | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (5):
- Placebo - Confirmatory Phase (Placebo Comparator): Participants received donepezil matched placebo tablets orally, once daily for 12 weeks in the confirmatory phase.
  Interventions: Drug: Donepezil matched placebo
- Donepezil 5 mg - Confirmatory Phase (Experimental): Participants received donepezil tablets orally, once daily for 12 weeks. Treatment began with 3 mg for 2 weeks, and then the dose was increased to 5 mg for 10 weeks in the confirmatory phase.
  Interventions: Drug: Donepezil 5 mg
- Donepezil 10 mg - Confirmatory Phase (Experimental): Participants received donepezil tablets orally, once daily for 12 weeks. Treatment began with 3 mg for 2 weeks, and then the dose was increased to 5 mg for 4 weeks. Thereafter, the dose was increased to 10 mg for 6 weeks in the confirmatory phase.
  Interventions: Drug: Donepezil 10 mg
- Placebo to Donepezil (5 +10 mg) - Extension Phase (Experimental): Participants previously receiving donepezil matched placebo up to Week 12 in the Confirmatory Phase, continued placebo until Week 16 (at the beginning of the Extension Phase). Participants received 3 mg of donepezil, and the dose was then increased to 5 mg at Week 18 and to 10 mg at Week 24. After Week 24, dose reduction to 5 mg was allowed if continuation at 10 mg caused any safety concerns.
  Interventions: Drug: Donepezil 10 mg
- Donepezil (5 +10 mg) - Extension Phase (Experimental): Participants previously receiving donepezil (5 mg or 10 mg) up to Week 12 in the Confirmatory Phase, maintained allocated treatment and dosages until Week 24. In the 5 mg group of the Confirmatory Phase, the dose was increased to 10 mg at Week 24. After Week 24, dose reduction to 5 mg was allowed if continuation at 10 mg caused any safety concerns.
  Interventions: Drug: Donepezil 10 mg

INTERVENTIONS:
Drug: Donepezil 5 mg — Donepezil tablets orally, once daily, uptitrated from 3 to 5 mg
  Other Names: E2020
  Arms: Donepezil 5 mg - Confirmatory Phase
Drug: Donepezil 10 mg — Donepezil tablets orally, once daily, uptitrated from 3 to 5 mg and then the dose was increased to 10 mg
  Other Names: E2020
  Arms: Donepezil (5 +10 mg) - Extension Phase; Donepezil 10 mg - Confirmatory Phase; Placebo to Donepezil (5 +10 mg) - Extension Phase
Drug: Donepezil matched placebo
  Arms: Placebo - Confirmatory Phase

SUMMARY:
The purpose of this study is to confirm the efficacy of E2020 in patients with dementia with Lewy bodies (DLB).

DETAILED DESCRIPTION:
This 52-week study consisted of 16-week randomized placebo-controlled (RCT, including 12-week Confirmatory Phase) and 36-week open-label extension phases. Of 142 DLB patients enrolled in the RCT phase (three arms: placebo, 5 mg, and 10 mg), 110 entered the extension phase. The placebo group of the RCT phase initiated active treatment at week 16, and the active groups maintained allocated treatment and dosages until week 24. After week 24, all patients received 10 mg. Dose reduction to 5 mg for safety concerns was allowed.

ELIGIBILITY:
Inclusion Criteria

1. Patients diagnosed as probable dementia with Lewy bodies (DLB) according to the consensus diagnostic criteria for DLB
2. Patients having caregivers throughout the study who submited written consent to cooperate with this study, who routinely stayed with patients 3 days or more a week (at least 4 hours a day), provided patients' information necessary for this study, assisted treatment compliance, and escorted the patients on required visits to study institution
3. Clinical Dementia Rating (CDR) score ≥ 0.5
4. Mini-Mental State Examination (MMSE) score of 10 to 26

Exclusion Criteria

1. Patients diagnosed with Parkinson's disease with dementia (PDD)
2. Patients who received anti-dementia drug therapy at the same institution
3. Patients who received anti-dementia drug therapy within 12 weeks before start of Screening
4. Patients with a complication of serious neuropsychiatric disease(s) such as stroke, brain tumor, schizophrenia, epilepsy, normal pressure hydrocephalus, mental retardation, brain trauma with unconsciousness, or a history of brain surgery causing unrecovered deficiency
5. Patients with severe extrapyramidal disorders (Hoehn and Hahr staging score ≥ IV)
6. Patients whose systolic blood pressure was less than 90 mmHg or pulse rate was less than 50 bpm at screening

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2011-02; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masaki Nakagawa, Study Director — Neuroscience Clinical Development Section. JAC PCU
Locations (56):
- Japan (56):
  - Anjo-shi, Aichi-ken
  - Nagoya, Aichi-ken
  - Toyokawa-shi, Aichi-ken
  - Chiba, Chiba
  - Fukui-shi, Fukui
  - Yoshida-gun, Fukui
  - Fukuoka, Fukuoka
  - Kitakyushu-shi, Fukuoka
  - Omuta-shi, Fukuoka
  - Gifu, Gifu
  - Mizunami-shi, Gifu
  - Fujioka-shi, Gunma
  - Maebashi, Gunma
  - Kure-shi, Hiroshima
  - Miyoshi-shi, Hiroshima
  - Otake-shi, Hiroshima
  - Obihiro-shi, Hokkaido
  - Sapporo, Hokkaido
  - Himeji-shi, Hyōgo
  - Kobe, Hyōgo
  - Yabu-shi, Hyōgo
  - Bando-shi, Ibaraki
  - Hitachi-shi, Ibaraki
  - Kahoku, Ishikawa-ken
  - Morioka, Iwate
  - Fujisawa-shi, Kanagawa
  - Kochi, Kochi
  - Koshi-shi, Kumamoto
  - Kumamoto, Kumamoto
  - Kyoto, Kyoto
  - Uji-shi, Kyoto
  - Sendai, Miyagi
  - Higashimorokata-gun, Miyazaki
  - Ina-shi, Nagano
  - Kitaazumi-gun, Nagano
  - Matsumoto-shi, Nagano
  - Nishisonogi-gun, Nagasaki
  - Nagaoka-shi, Niigata
  - Sanjo-shi, Niigata
  - Tsubame-shi, Niigata
  - Yufu-shi, Oita Prefecture
  - Osaka, Osaka
  - Sakai-shi, Osaka
  - Sennan-shi, Osaka
  - Suita-shi, Osaka
  - Ageo-shi, Saitama
  - Kasukabe-shi, Saitama
  - Saitama-shi, Saitama
  - Fuji-shi, Shizuoka
  - Hamamatsu, Shizuoka
  - Shizuoka, Shizuoka
  - Koto-ku, Tokyo
  - Ōta-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Suginami-ku, Tokyo

REFERENCES:
- [Derived] Mori E, Ikeda M, Nagai R, Matsuo K, Nakagawa M, Kosaka K. Long-term donepezil use for dementia with Lewy bodies: results from an open-label extension of Phase III trial. Alzheimers Res Ther. 2015 Feb 3;7(1):5. doi: 10.1186/s13195-014-0081-2. eCollection 2015. PMID 25713600
- [Derived] Ikeda M, Mori E, Matsuo K, Nakagawa M, Kosaka K. Donepezil for dementia with Lewy bodies: a randomized, placebo-controlled, confirmatory phase III trial. Alzheimers Res Ther. 2015 Feb 3;7(1):4. doi: 10.1186/s13195-014-0083-0. eCollection 2015. PMID 25713599

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the 'Placebo to Donepezil (5+10 mg) Extension Phase' arm, 37 of 46 participants started active treatment at Week 16.
Period: Confirmatory Phase
Arm/Group | Placebo - Confirmatory Phase | Donepezil 5 mg - Confirmatory Phase | Donepezil 10 mg - Confirmatory Phase | Placebo to Donepezil (5 +10 mg) - Extension Phase | Donepezil (5 +10 mg) - Extension Phase
Started | 46 | 47 | 49 | 0 | 0
Completed | 37 | 31 | 43 | 0 | 0
Not Completed | 9 | 16 | 6 | 0 | 0
Not completed — Adverse Event | 5 | 10 | 1 | 0 | 0
Not completed — Participant's Choice | 3 | 5 | 3 | 0 | 0
Not completed — Other | 1 | 1 | 2 | 0 | 0
Period: Extension Phase
Arm/Group | Placebo - Confirmatory Phase | Donepezil 5 mg - Confirmatory Phase | Donepezil 10 mg - Confirmatory Phase | Placebo to Donepezil (5 +10 mg) - Extension Phase | Donepezil (5 +10 mg) - Extension Phase
Started | 0 | 0 | 0 | 46 | 96
Completed | 0 | 0 | 0 | 34 | 66
Not Completed | 0 | 0 | 0 | 12 | 30
Not completed — Adverse Event | 0 | 0 | 0 | 7 | 16
Not completed — Participant's Choice | 0 | 0 | 0 | 4 | 11
Not completed — Other | 0 | 0 | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Population: The data is based on Full Analysis Set, defined as all the randomized patients who received the study drug at least once and had valid efficacy assessment data at more than one point.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo - Confirmatory Phase | Donepezil 5 mg - Confirmatory Phase | Donepezil 10 mg - Confirmatory Phase | Total
Number analyzed (Participants) | 44 | 45 | 49 | 138
Age, Continuous [Mean (Standard Deviation); unit: Years] | 77.2 (6.1) | 78.8 (5.1) | 77.7 (6.8) | 77.9 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 28 | 80
  Male | 17 | 20 | 21 | 58
Mini-Mental State Examination (MMSE) Score [Mean (Standard Deviation); unit: Unit on a scale] — The score ranged from 0 to 30, with a higher score indicating better function.
  Unit on a scale | 20.3 (4.2) | 20.6 (4.1) | 20.3 (4.8) | 20.4 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mini-Mental State Examination (MMSE) Score
Description: The MMSE was used to measure cognitive impairment. The MMSE can evaluate overall cognitive function, and is widely used for the assessment of cognitive impairment in dementia patients. The questionnaire consists of 11 items, and each item aims to evaluate different cognitive domains such as orientation, memory, attention, and construction. The score ranged from 0 to 30, with a higher score indicating better function. A positive change score indicated improvement from baseline. Data are presented as change from baseline in mean MMSE +/- standard deviation.
Time Frame: Week 12 for Confirmatory Phase
Population: Full Analysis Set: Efficacy was analyzed in the full analysis set, including the randomized participants who received the study drug at least once and had valid efficacy assessment data at more than one point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo - Confirmatory Phase | Donepezil 5 mg - Confirmatory Phase | Donepezil 10 mg - Confirmatory Phase
Number analyzed (Participants) | 44 | 43 | 49
Units on a scale | 0.6 (3.0) | 1.4 (3.4) | 2.2 (2.9)

2. Primary Outcome: Change From Baseline in Neuropsychiatric Inventory (NPI-2) Score
Description: The NPI was a questionnaire that quantified psychiatric symptoms and behavioral disorders in dementia. A total of 12 items (the original NPI-10 consisting of 10 behavioral domains: delusions, hallucinations, agitation/aggression, dysphoria, anxiety, euphoria, apathy, disinhibition, irritability/lability, and aberrant motor behavior, supplemented by 2 dementia with Lewy bodies (DLB)-relevant domains of sleep, and cognitive fluctuation [reported as cognitive fluctuation inventory]) were assessed. The score of each item was calculated as frequency (scale: 1=occasionally to 4=very frequently) x Severity (scale: 1=Mild to 3=Severe). The NPI-2 was calculated as the sum of the scores for hallucinations and cognitive fluctuation, to yield a possible total score of 0 to 24. Lower score=less severity. A negative change score from baseline indicated improvement. Data are presented as change from baseline in mean NPI-2 +/- standard deviation.
Time Frame: Week 12 for Confirmatory Phase
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo - Confirmatory Phase | Donepezil 5 mg - Confirmatory Phase | Donepezil 10 mg - Confirmatory Phase
Number analyzed (Participants) | 44 | 45 | 49
Units on a scale | -2.0 (4.2) | -1.7 (4.3) | -2.9 (4.7)

ADVERSE EVENTS:
Time Frame: For each patient from first dose of study drug administration up to 30 days from last dose of study drug or up to approximately Week 12 for Confirmatory Phase and Week 52 for Extension Phase
Description: Safety Analysis Set: The safety analysis set comprised of all patients who received at least one dose and had a postbaseline safety assessment. In the 'Placebo to Donepezil (5+10 mg) Extension Phase' arm, 37 of 46 participants started active treatment at Week 16.
Arm/Group | Placebo - Confirmatory Phase | Donepezil 5 mg - Confirmatory Phase | Donepezil 10 mg - Confirmatory Phase | Placebo to Donepezil (5 +10 mg) - Extension Phase | Donepezil (5 +10 mg) - Extension Phase
Serious Adverse Events (participants affected / at risk) | 5/46 | 4/47 | 1/49 | 9/37 | 12/96
Other Adverse Events (participants affected / at risk) | 23/46 | 18/47 | 17/49 | 31/37 | 62/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - Confirmatory Phase (N=46) | Donepezil 5 mg - Confirmatory Phase (N=47) | Donepezil 10 mg - Confirmatory Phase (N=49) | Placebo to Donepezil (5 +10 mg) - Extension Phase (N=37) | Donepezil (5 +10 mg) - Extension Phase (N=96)
Hypertension (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0
Decreased appetite (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Paranoia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - Confirmatory Phase (N=46) | Donepezil 5 mg - Confirmatory Phase (N=47) | Donepezil 10 mg - Confirmatory Phase (N=49) | Placebo to Donepezil (5 +10 mg) - Extension Phase (N=37) | Donepezil (5 +10 mg) - Extension Phase (N=96)
Pyrexia (General disorders) | 0 | 0 | 3 | 0 | 3
Nasopharyngitis (Infections and infestations) | 7 | 4 | 2 | 18 | 17
Contusion (Injury, poisoning and procedural complications) | 4 | 0 | 1 | 6 | 7
Pollakiuria (Renal and urinary disorders) | 0 | 3 | 0 | 0 | 3
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 2 | 2
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1 | 4 | 6
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 5
Nausea (Gastrointestinal disorders) | 1 | 2 | 1 | 3 | 4
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 2
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0 | 0 | 3 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 2 | 0
Glucose urine present (Investigations) | 0 | 0 | 1 | 1 | 5
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 2 | 0 | 5
Weight decreased (Investigations) | 2 | 1 | 0 | 2 | 2
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 2 | 2 | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 2 | 5
Parkinsonism (Nervous system disorders) | 2 | 2 | 4 | 5 | 12
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 3 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Agitation (Psychiatric disorders) | 2 | 1 | 0 | 2 | 3
Insomnia (Psychiatric disorders) | 0 | 2 | 0 | 0 | 5
Sleep disorder (Psychiatric disorders) | 2 | 1 | 0 | 3 | 1
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2 | 2
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2 | 1
Irritability (General disorders) | 1 | 1 | 0 | 2 | 2
Oedema peripheral (General disorders) | 0 | 0 | 0 | 2 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other